CLINICAL TRIAL: NCT02557906
Title: Prospective, Multi-centre, Observational Trial Evaluating Outcomes of Immediate Breast Reconstruction Using an Implant and Acellular Dermal Matrix (SurgiMend) or Autologous Tissue
Brief Title: Evaluating Outcomes of Immediate Breast Reconstruction (POBRAD-M)
Acronym: POBRAD-M
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 153962
Record Dates: First submitted 2015-07-28; First posted 2015-09-23 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Breast Neoplasms; Breast Diseases
Keywords: Acellular dermal matrix; ADM; SurgiMend; Breast reconstruction; Immediate breast reconstruction; Autologous reconstruction; Biological mesh
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases | interventions — Mammaplasty; Surgimend

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Implant and Surgimend (Experimental): Breast reconstruction surgery with an implant and an ADM (Surgimend)
  Interventions: Procedure: Breast reconstruction - implant and an ADM (SurgiMend)
- Autologous tissue (Active Comparator): Breast reconstruction surgery with autologous tissue
  Interventions: Procedure: Breast reconstruction- autologous tissue
- Implant + dermal sling/LD flap (Active Comparator): Breast reconstruction surgery using a dermal sling or a latissimus dorsi (LD)flap
  Interventions: Procedure: Breast reconstruction- implant + dermal sling/LD flap

INTERVENTIONS:
Procedure: Breast reconstruction - implant and an ADM (SurgiMend) — Skin or nipple sparing mastectomy and immediate breast reconstruction with implants and SurgiMend
  Other Names: SurgiMend
  Arms: Implant and Surgimend
Procedure: Breast reconstruction- autologous tissue — Skin or nipple sparing mastectomy and immediate breast reconstruction with autologous tissue
  Arms: Autologous tissue
Procedure: Breast reconstruction- implant + dermal sling/LD flap — Skin or nipple sparing mastectomy and immediate breast reconstruction using an implant and a dermal sling or a latissimus dorsi flap
  Arms: Implant + dermal sling/LD flap

SUMMARY:
Some women with breast cancer have their whole breast removed as part of their treatment (mastectomy). Of these women, around 31% have more surgery to create a new breast.There are two main ways to create a new breast(i)using tissue from elsewhere on the body ("autologous" reconstruction )or (ii)using a silicone implant.

In recent years, it has been reported that by using a material called an "acellular dermal matrix" (ADM) the results of breast reconstruction surgery using an implant can be improved. ADMs are materials which originally come from animal or human skin. They act like a sling, supporting the lower part of an implant beneath the skin.

Although ADMs have been approved for used in breast reconstruction and are safe, there is very little high quality evidence to back up their reported benefits, and some studies have suggested their use may in fact increase complications.

The main purpose of this study is to find out what the actual risks and benefits of using an ADM in breast reconstruction surgery are. The investigators will follow the progress of women who have an implant based reconstruction to observe if participants develop problems; what those problems are and how participants feel about the results of their surgery. The investigators also follow the progress of women who undergo autologous reconstruction or alternative reconstructive techniques using an implant for the same reasons.

DETAILED DESCRIPTION:
Despite the widespread adoption of acellular dermal matrices (ADMs) in breast reconstruction, there is limited prospective or high quality evidence on the outcomes of their use. The majority of studies on ADM are poor quality retrospective cohort studies with ill-defined, non-standardised outcome measures and heterogeneous patient populations. Recent systematic reviews have raised concerns of increased infection and seroma rates associated with ADM use which, if correct, may negate their reported advantages. Furthermore there is little high quality evidence to confirm the benefits associated with their use such as improved aesthetic outcomes.

The POBRAD-M is a prospective, multicentre trial which will evaluate the early and late outcomes of immediate breast reconstruction using either an implant and ADM, autologous tissue or an alternative implant-based technique. All participants must have been deemed suitable at the outset for implant based reconstruction with an ADM irrespective of their final procedure choice. All participants will be followed up at 30 days, 3 months and 12 months to record the incidence of complications (to include implant loss, infection, seroma, haematoma and skin necrosis). Additionally Patient Reported Outcomes measures using the BREAST-Q questionnaire will be determined at 30 days and 12 months, and aesthetic outcome will be determined by panel assessment of post-operative photographs at 12 months post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent given
* Unilateral or bilateral mastectomy (therapeutic, contra lateral or prophylactic)
* Immediate reconstruction;
* Suitable for immediate implant reconstruction with ADM

Exclusion Criteria:

* Patients unable to provide informed consent to participate in trial
* Patients unavailable for follow-up
* Not eligible for immediate breast reconstruction using an ADM

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2014-07; Primary Completion 2016-01 (Actual); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events | 30 days
  Adverse events defined as implant loss, infection, haematoma, seroma, skin necrosis in all cohorts
Number of patients with adverse events | 3 months
  Adverse events defined as implant loss, infection, haematoma, seroma, skin necrosis in all cohorts
Number of patients with adverse events | 12 months
  Adverse events defined as implant loss, infection, haematoma, seroma, skin necrosis in all cohorts

SECONDARY OUTCOMES:
Aesthetic outcome measured by Photographic assessment | 12 months
  Photographic assessment
BREAST-Q questionnaire score | 30 days
  Patient-reported outcome measures using the BREASTQ questionnaire
BREAST-Q questionnaire score | 12 months
  Patient-reported outcome measures using the BREASTQ questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Michael Douek, MD FRCS, Principal Investigator — King's College London
Locations (6):
- United Kingdom (6):
  - Royal Hampshire County Hospital, Winchester, Hampshire
  - Frimley Park Hospitals NHS Foundation Trust, Frimley
  - Leeds Teaching Hospitals, Leeds
  - Department of Research Oncology, King's College London, London
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - Royal Cornwall Hospital, Truro